CLINICAL TRIAL: NCT03926013
Title: A Phase 1, First-in-Human, Dose Escalation Study of JNJ-63898081, in Subjects With Advanced Stage Solid Tumors
Brief Title: A Study of JNJ-63898081 in Participants With Advanced Stage Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108593; 63898081EDI1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-04-22; First posted 2019-04-24 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): Participants with metastatic castration-resistant prostate cancer (mCRPC) will receive JNJ-63898081. Ascending dose levels will be sequentially tested.
  Interventions: Drug: JNJ-63898081
- Part 2: Dose Expansion (Experimental): Participants with mCRPC or renal cell carcinoma (RCC) will receive JNJ-63898081 at the recommended Phase 2 dose (RP2D) determined in Part 1.
  Interventions: Drug: JNJ-63898081

INTERVENTIONS:
Drug: JNJ-63898081 — JNJ-63898081 will be administered.

SUMMARY:
The main purpose of this study are to determine the recommended Phase 2 dose (RP2D) regimen and the maximum tolerated dose, and to determine the safety of JNJ-63898081.

ELIGIBILITY:
Inclusion Criteria:

* Histology: Part 1: Metastatic castration-resistant prostate cancer (mCRPC) with histologic confirmation of adenocarcinoma. Adenocarcinoma with small-cell or neuroendocrine features is allowed. mCRPC is defined by prostate Cancer Working Group (PCWG )3 criteria. Part 2: mCRPC as defined above or pathologically confirmed metastatic renal cell carcinoma (RCC) as defined by world health organization (WHO) 2016 Classifications
* Measurable or evaluable disease: Part 1: Either measurable or evaluable disease for prostate cancer. Part 2: At least one measurable lesion as per RECIST v1.1.
* Evidence of disease progression on prior therapy that requires a new line of treatment
* Participants with accessible lesions enrolled in selected pharmacokinetic (PK)/pharmacodynamics (PD) cohorts and in Part 2 must agree to undergo the mandatory fresh tumor biopsies, unless collection of the biopsy presents a safety risk

Exclusion Criteria:

* Less than 2 weeks between prior anticancer treatment (including radiotherapy) discontinuation and the first dose of study drug, and toxicities have not returned to Grade less than or equal to (<=) 1 or baseline
* Prior treatment with prostate-specific membrane antigen (PSMA)-targeted therapy except for PSMA-targeted vaccine is permitted
* Solid organ or bone marrow transplantation
* Seizure or known condition that may predispose to seizure or intracranial masses
* Other active malignancy requiring systemic treatment <=12 months prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-09-02 (Actual)

PRIMARY OUTCOMES:
Part 1 and Part 2: Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Approximately 3 years
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Part 1: Number of Participants with Dose-Limiting Toxicity (DLT) | Approximately 3 years
  Number of participants with DLT will be assessed. The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity.
Part 1: Severity of Adverse Events as Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) | Approximately 3 years
  Severity of AEs has 5 grades based on CTCAE criteria: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening consequences; Grade 5: Death.

SECONDARY OUTCOMES:
Part 1 and Part 2: Serum Concentrations of JNJ-63898081 | Approximately 3 years
  Serum samples will be analyzed to determine concentrations of JNJ-63898081 using a validated method.
Part 1 and 2: Systemic Cytokine Concentrations | Approximately 3 years
  A panel of cytokines, including those proinflammatory ones, will be measured.
Part 1 and 2: Number of Participants with JNJ-63898081 Antibodies | Approximately 3 years
  Anti-JNJ-63898081 antibodies will be evaluated in serum samples collected from all participants.
Serum Prostate Specific Antigen (PSA) Concentration | Approximately 3 years
  Serum prostate specific antigen (PSA) concentration will be assessed.
Objective Response Rate (ORR) | Approximately 3 years
  ORR is defined as the proportion of participants who have a PR or better according to the disease-specific response criteria. Evaluation of prostate treatment response will be performed according to Prostate Cancer Working Group 3 (PCWG3).
Duration of Response | Approximately 3 years
  Duration of response (DOR) will be calculated from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in the disease-specific response criteria, or death due to any cause, whichever occurs first. Evaluation of prostate treatment response will be performed according to Prostate Cancer Working Group 3 (PCWG3).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (7):
- United States (5):
  - University of California, San Francisco, San Francisco, California
  - NIH Clinical Center, Bethesda, Maryland
  - Columbia University Medical Center, New York, New York
  - University of Utah, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
- Canada (2):
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency